CLINICAL TRIAL: NCT03019731
Title: Behavioral Therapy for Tourette Syndrome: Home-Based and Therapist-Administered
Brief Title: Behavioral Therapy for Tourette Syndrome
Acronym: BTTS:HBTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Tourette Association of America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00111766
Record Dates: First submitted 2016-12-14; First posted 2017-01-13 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2019-09

CONDITIONS: Tourette Syndrome
Keywords: Tics; Behavioral therapy; Neurologic Examination
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with Tourette syndrome (Experimental): Eligible children, between ages 7-13 years, with the diagnosis of Tourette syndrome or chronic motor/vocal tic disorder will be recruited from the Tourette Syndrome Clinics at Johns Hopkins (Dr. Singer). The Johns Hopkins Center has been acclaimed a Center of Excellence by the Tourette Association of America. This center currently follows more than 1,000 tic patients and averages 4-6 new referrals and 4 follow up patients weekly. Children will be randomly assigned to either the Therapist-directed Behavioral Therapy group or the Home-based DVD therapy group.
  Interventions: Behavioral: Therapist-directed Behavioral Therapy; Behavioral: Home-based DVD Therapy

INTERVENTIONS:
Behavioral: Therapist-directed Behavioral Therapy — The therapist-directed behavioral therapy group will have their first appointment scheduled within one week of assignment. In the Therapist-directed face-face training program, training instructions will be manualized, in order to match the parent instructional guidelines provided in the home-based DVD. This manual will include the specific psychoeducation, awareness training, competing response training, differential reinforcement of incompatible behaviors, and other adaptive behavioral instructions contained within the home-based DVD. The therapist will match the sequence and required components within the behavior-based training DVD. Face-face training will be administered across 10 weeks (6 weekly sessions followed by 2 bi-weekly sessions).
Behavioral: Home-based DVD Therapy — In order to mimic the slight delay between randomization and start of the therapist-directed treatment, those assigned to the Home-based DVD cohort will have the DVD and training materials mailed to their homes. Parents will also receive a written instructional form and a log sheet for tracking the use of the DVD and the time and duration of practice sessions. Any questions regarding patient care and treatment will be directed to Dr. Singer.

SUMMARY:
This research is being done to determine whether a home-based behavioral therapy can be successfully used to treat tics in children with Tourette syndrome (TS). Behavioral therapy administered by a trained therapist has been shown to be helpful in reducing tics in children with Tourette syndrome. In this study, the investigators want to determine whether an instructional video can provide parents of children with TS with the tools necessary to successfully use behavioral therapy at home. The investigators also want to determine the effectiveness of home-based behavioral therapy as compared to improvement achieved when the therapy is provided by a trained therapist.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a neurodevelopmental disorder with childhood onset characterized by the presence of chronic motor and vocal (phonic) tics. Tics typically begin between the ages of 4 - 7 years, frequently persist, and often lead to psychosocial, physical, functional, and academic difficulties. Epidemiological studies have shown that about 20-30% of children exhibit tics in a classroom setting whereas the estimated prevalence of impairing cases of TS is 1/100 - 1/1000 individuals. There is no cure for tics and a variety of behavioral and pharmacotherapies have been used successfully to suppress tics. Comprehensive Behavioral Intervention for Tics (CBIT) has been shown to be beneficial in several large trials as has habit reversal training (HRT), one of its major components. In the past, it has been suggested that only "competent and trained practitioners should administer CBIT." This proposal challenges that concept and believes that one can establish a successful front-line home-based CBIT treatment program that would be beneficial for the treatment of patients with tic symptoms throughout the country.

CBIT is a safe, effective, front-line treatment for TS. Nevertheless, the investigators emphasize the acute shortage of appropriately trained clinicians available to assist affected individuals. Hence, in this proposal the investigators will assess the effectiveness of a behavioral home-based, parent administered treatment by investigating at Johns Hopkins Hospital whether the home-based digital video disc (DVD) reduces tic severity comparable to that achieved with face-to-face treatment administered by an experienced therapist. The investigators' confidence in the success of this project is based on prior experiences with another childhood movement disorder, primary complex motor stereotypies. The potential significance of this project is enormous, recognizing that home-based therapy reduces health care costs, visits to practitioners, the need to train large numbers of therapists, and most importantly provides direct, available care for a greater number individuals affected with tics.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for TS or a chronic motor/vocal tic disorder (CTD). TS as defined by the TS Classification Study Group, includes onset before 18 years, multiple involuntary motor tics, one or more vocal tics, a waxing and waning course, the gradual replacement of old symptoms with new ones, the presence of tics for more than one year, the absence of other medical explanations for tics, and the observation of tics by a reliable examiner. CTD, criteria are as above, except that only motor or vocal tics are required
* Age 7-13 years, either gender
* Observable tics, achieving a minimum score > 20 for TS or > 15 for CTD on the Total Tic Severity score of the Yale Global Tic Severity Scale (YGTSS)
* Tic symptoms must be severe enough to warrant therapy; [e] Tics are not controlled with current medication or individuals are tic-suppressing drug naïve
* The concurrent use of other tic-suppressing medications will be permitted, if the subject has been on a stable dose for more than six weeks and agrees to maintain a constant dosage throughout the study; [6] The concurrent use of medication for Attention-Deficit Hyperactivity Disorder (ADHD) or Obsessive Compulsive Disorder (OCD) is also permitted if the participant has been on a stable dose for more than six weeks and agrees to maintain a constant dosage throughout the study.

Participants will be included in the study if they have had less than four previous sessions of habit reversal training. The investigators will not allow the study to interfere with simultaneous behavioral treatment. In this study, the investigators will assess whether caregiver-directed behavioral therapy using an instructional DVD will help patients who would like behavioral therapy, but the patients do not live close enough to Johns Hopkins for frequent visits.

Exclusion Criteria:

* Secondary tics
* Significant medical illness or a chronic neurological condition (i.e., seizure disorder, developmental neurological conditions, acquired brain injuries
* Current major depression, generalized anxiety disorder, separation anxiety disorder, psychotic symptoms (based upon clinical evaluation), pervasive developmental disorder, autism, intellectual disability (I.Q. less than 70), anorexia/bulimia, or substance abuse
* Individuals with significant OCD, not controlled by medication, will be excluded
* Four or more previous sessions of habit reversal training.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
The Yale Global Tic Severity Scale Total Tic Score (TTS) | Baseline (0 weeks)
  The YGTSS is a clinician-rated measure that begins with the completion of a checklist of all tics present in the past week. Current motor and vocal tics are then rated on 5 dimensions each on a 0-5 scale: tic number, frequency, duration, intensity, and complexity. Each of the dimensions is scored separately for motor and vocal tics and summed to yield separate motor and vocal tic subscale scores (range 0-25). These subscales are then combined to produce a total tic severity score (range 0-50). An associated impairment scale (range 0-50) assesses tic-related disability during the past week. The YGTSS has demonstrated acceptable internal consistency and acceptable convergent and divergent validity.

SECONDARY OUTCOMES:
Clinical Global Impressions-Improvement scale (CGI) | Baseline (0 weeks)
  The Clinical Global Impressions-Improvement scale (CGI-I) is a clinician rating to assess overall clinical improvement based on observed and patient-reported symptom severity and symptom-related impairment. Scores range from 1 to 7 where: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. Responders are defined as those who receive a score of 1 or 2 on the CGI-I.

OTHER OUTCOMES:
Parent Tic Questionnaire (PTQ) | Baseline (0 weeks)
  The Parent Tic Questionnaire (PTQ) measures the number, frequency, intensity of motor and vocal tics. For each tic endorsed in a checklist of common motor and vocal tics over the past week, the parent rates its frequency (4 = constantly, 3 = hourly, 2 = daily, 1 = weekly, 0 = absent) and intensity or noticeable (1-4). An overall score is computed by summing the motor and vocal tic subscale scores. The PTQ has been shown to have excellent internal consistency and test-retest reliability.
The Yale Global Tic Severity Scale Total Tic Score (TTS) | At 5 weeks
  The YGTSS is a clinician-rated measure that begins with the completion of a checklist of all tics present in the past week. Current motor and vocal tics are then rated on 5 dimensions each on a 0-5 scale: tic number, frequency, duration, intensity, and complexity. Each of the dimensions is scored separately for motor and vocal tics and summed to yield separate motor and vocal tic subscale scores (range 0-25). These subscales are then combined to produce a total tic severity score (range 0-50). An associated impairment scale (range 0-50) assesses tic-related disability during the past week. The YGTSS has demonstrated acceptable internal consistency and acceptable convergent and divergent validity.
Clinical Global Impressions-Improvement scale (CGI) | At 5 weeks
  The Clinical Global Impressions-Improvement scale (CGI-I) is a clinician rating to assess overall clinical improvement based on observed and patient-reported symptom severity and symptom-related impairment. Scores range from 1 to 7 where: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. Responders are defined as those who receive a score of 1 or 2 on the CGI-I.
Parent Tic Questionnaire (PTQ) | At 5 weeks
  The Parent Tic Questionnaire (PTQ) measures the number, frequency, intensity of motor and vocal tics. For each tic endorsed in a checklist of common motor and vocal tics over the past week, the parent rates its frequency (4 = constantly, 3 = hourly, 2 = daily, 1 = weekly, 0 = absent) and intensity or noticeable (1-4). An overall score is computed by summing the motor and vocal tic subscale scores. The PTQ has been shown to have excellent internal consistency and test-retest reliability.
The Yale Global Tic Severity Scale Total Tic Score (TTS) | At 10 weeks
  The YGTSS is a clinician-rated measure that begins with the completion of a checklist of all tics present in the past week. Current motor and vocal tics are then rated on 5 dimensions each on a 0-5 scale: tic number, frequency, duration, intensity, and complexity. Each of the dimensions is scored separately for motor and vocal tics and summed to yield separate motor and vocal tic subscale scores (range 0-25). These subscales are then combined to produce a total tic severity score (range 0-50). An associated impairment scale (range 0-50) assesses tic-related disability during the past week. The YGTSS has demonstrated acceptable internal consistency and acceptable convergent and divergent validity.
Clinical Global Impressions-Improvement scale (CGI) | At 10 weeks
  The Clinical Global Impressions-Improvement scale (CGI-I) is a clinician rating to assess overall clinical improvement based on observed and patient-reported symptom severity and symptom-related impairment. Scores range from 1 to 7 where: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. Responders are defined as those who receive a score of 1 or 2 on the CGI-I.
Parent Tic Questionnaire (PTQ) | At 10 weeks
  The Parent Tic Questionnaire (PTQ) measures the number, frequency, intensity of motor and vocal tics. For each tic endorsed in a checklist of common motor and vocal tics over the past week, the parent rates its frequency (4 = constantly, 3 = hourly, 2 = daily, 1 = weekly, 0 = absent) and intensity or noticeable (1-4). An overall score is computed by summing the motor and vocal tic subscale scores. The PTQ has been shown to have excellent internal consistency and test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Singer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No